CLINICAL TRIAL: NCT06605872
Title: An Open, Multicentre, Prospective, Non-interventional Study of the CE-marked Medical Device GlucoTab, According to Intended Use Without Additional Invasive and Stressful Measures With a Matched Retrospective Control Group
Brief Title: DigiDiab Pilot: Impact Study Hospital
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 230206 EITHealth-hospital
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: GlucoTab; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GlucoTab Prospective Group
  Interventions: Device: GlucoTab
- Retrospective control group
  Interventions: Other: Diabetes Treatment

INTERVENTIONS:
Device: GlucoTab — Insulin therapy will be started and adjusted according to the GlucoTab system with incorporated software algorithm. Insulin therapy prescription for the next 24 hours is suggested once daily by the GlucoTab system taking previous insulin doses, glucose readings, patient age, renal function and insulin sensitivity into account. The goal of the algorithm is to maintain fasting and premeal glucose concentrations between 100-140 mg/dl, (5.6 to 7.8 mmol/l).
  Groups: GlucoTab Prospective Group
Other: Diabetes Treatment — Diabetes Standard Care
  Groups: Retrospective control group

SUMMARY:
GlucoTab is an innovative workflow and decision support tool for standardised diabetes management by healthcare professionals which provides automated and personalised dosage recommendations for different insulin therapy regimens.

DETAILED DESCRIPTION:
GlucoTab has already been tested in several clinical trials in Austria and has consecutively obtained the CE-mark that is valid throughout European countries.

The current study aims to further develop, implement and evaluate GlucoTab in different European pilot regions. For this reason, GlucoTab will be translated in different languages and tested in Sweden, Denmark, and Spain.

ELIGIBILITY:
Inclusion Criteria:

* informed consent obtained after being advised of the nature of the study
* a documented history of type 2 diabetes prior to inclusion or new-onset hyperglycaemia which requires s.c. insulin therapy during hospital stay
* admission to either surgical or internal medicine ward
* an expected length of hospital stay for at least 48 hours after enrolment

Exclusion Criteria:

* type 1 diabetes mellitus
* intravenous insulin therapy
* hyperglycaemic episodes (ketoacidosis, hyperosmolar state) if they require intravenous insulin therapy
* continuous subcutaneous insulin infusion
* gestational diabetes or pregnancy
* known or suspected allergy to insulin
* total parenteral nutrition
* any mental condition rendering the patient incapable of giving his/her consent
* any disease or condition which according to the investigator or treating physician would interfere with the trial or the safety of the patient

Inclusion and exclusion criteria will be the same as above for the retrospective CG with the exception of:

* period of time will be from September 2022 to September 2023
* no informed consent will be obtained from the retrospective CG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are non-critically ill patients with type 2 diabetes at general hospital wards who require s.c. insulin therapy during hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy - mean percentage of blood glucose values in target range | ≥ 24 hours after start of therapy by using the GlucoTab system four times daily
  Efficacy is assessed by measuring the mean percentage of blood glucose values in the target range 100 to 140 mg/dl (5.6 to 7.8 mmol/l)

SECONDARY OUTCOMES:
Usability - adherence to suggestions of the GlucoTab system | from enrollment to the end of treatment with a maximum of 21 days
  adherence to suggestions of the GlucoTab system
Safety - number of hypoglycaemic events | from enrollment to the end of treatment with a maximum of 21 days
  Safety is assessed by the number of hypoglycaemic events
Efficacy - mean daily blood glucose | from enrollment to the end of treatment with a maximum of 21 days
  mean daily blood glucose

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Joan XXIII de Tarragona, Tarragona, Spain